CLINICAL TRIAL: NCT06443333
Title: National, Multicentric Registry Study on Neuroimmunological Diseases in China
Acronym: NIDBase
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: XWZC20210115
Record Dates: First submitted 2024-05-10; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis; NMO Spectrum Disorder; Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease; Myasthenia Gravis; Autoimmune Encephalitis; Acute Disseminated Encephalomyelitis
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease; Myasthenia Gravis; Autoimmune Diseases of the Nervous System; Encephalomyelitis, Acute Disseminated | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — The biological samples of enrolled patients and healthy volunteers, such as blood and cerebrospinal fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neuroimmune diseases patient: Patients diagnosed with neuroimmune diseases by a neurologist.
  Interventions: Other: Data collection and follow-up observation
- Health Volunteers: Healthy adults undergoing medical examinations at the Xuanwu Hospital Physical Examination Center.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection and follow-up observation — At the time of enrollment, the patient's biological samples are collected to obtain genetic information. Following enrollment, trained investigators carry out a 2-year follow-up observation through face-to-face, telephone call or online visits. During the follow-up, basic clinical information, laboratory tests, imaging examinations, neurophysiology, clinical classification, medication use, and scale assessments are collected.
  Groups: neuroimmune diseases patient
Other: Data collection — Collect demographic and genetic information from healthy volunteers upon enrollment.
  Groups: Health Volunteers

SUMMARY:
The aim of this study is to establish a real-world clinical neuroimmune disease research cohort, to follow up and observe the prognosis of patients with different subtypes and subgroups, and to provide support for the treatment, early warning, and outcome prediction research of neuroimmune diseases.

DETAILED DESCRIPTION:
The purposes of this study are:(1)Establishing a clinical neuroimmune disease research cohort.(2)Collecting the blood, cerebrospinal fluid and other biological samples of the enrolled patients to discover and detect the new neural antibodies, so as to facilitate the diagnosis of related diseases.(3) Conducting in-depth exploration of the Genetic material of patients with neuroimmune diseases and healthy volunteers with second-generation sequencing technology, discovering the pathogenic genes and the mechanism of disease progression.The enrolled patients will be collected Clinical and therapeutic information. Blood and cerebrospinal fluid from the patients will be collected for sequencing analysis and antibody detection. They will also receive the 2-year follow-up with collection of basic clinical information, cognitive function, EDSS score, etc. Healthy volunteers will have their blood collected for sequencing analysis.

Finish the gene sequencing analysis of blood samples from enrolled patients and healthy volunteers to establish the disease gene database and the reference gene database of the healthy population and find the unique expression quantitative trait loci (eQTL) in China, so as to clarify the pathogenic genes and the key mechanism of neuroimmune disease occurrence and development.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed at Xuanwu Hospital, Capital Medical University with any of the following conditions:

  * Multiple Sclerosis (the criteria followed the Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria)
  * NMO Spectrum Disorder (the criteria followed the Diagnosis and Treatment Guidelines for Optic Neuromyelitis Spectrum Disorders in China 2016)
  * Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease (the criteria followed the Consensus of Chinese Experts on Diagnosis and Treatment of Anti-Myelin Oligodendrocyte Glycoprotein Immunoglobulin G Antibody-Associated Diseases)
  * Myasthenia Gravis (the criteria followed the Guidelines for the Diagnosis and Treatment of Myasthenia Gravis in China 2020)
  * Autoimmune Encephalitis (the criteria followed the China Expert Consensus on Diagnosis and Treatment of Autoimmune Encephalitis 2017)
  * Acute Disseminated Encephalomyelitis (the criteria are based on the article titled "Acute disseminated encephalomyelitis" 2007).
* Healthy adults who underwent a physical examination at the Physical Examination Center of Xuanwu Hospital, Capital Medical University

Exclusion Criteria:

* Women during pregnancy or lactation.
* Patients with other neurological diseases or serious mental diseases.
* Patients with serious liver and kidney function or other important organ dysfunction.
* Unable to cooperate with follow-up work and venous blood collection due to poor compliance of patients or healthy volunteers, or incomplete clinical and imaging data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients and healthy volunteers from China
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Annual recurrence rate | At 12 and 24 months after enrollment
  Whether there is recurrence in patients followed up at 12 and 24 months after enrollment

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale scores (EDSS) | At 6,12,18,24 months after enrollment
  Change from baseline in Expanded Disability Status Scale scores (EDSS，range from 0 to 10 points, with a higher score indicating a more severe degree of neurological impairment).
Change in MRI of head, optic nerve and spinal cord | At 6,12,18,24 months after enrollment
  whether there are New or enlarged lesions in T1WI, T2WI, T2 FLAIR, Sag bravo, DTI, and BOLD MRI of head, optic nerve and spinal cord in neuroimmune disease patients.
Change in serum and CSF autoimmune antibody status | At 6,12,18,24 months after enrollment
  Collect the patient's serum and cerebrospinal fluid to measure the types and concentrations of autoantibodies. Note any changes compared to the baseline.
Change in Activity of Daily Living Scale (ADL) | At 6,12,18,24 months after enrollment
  Change from baseline in Activity of Daily Living Scale (ADL, range from 14 to 56 points, with higher scores indicating poorer daily life abilities).
Change in the relative power spectral density | At 6,12,18,24 months after enrollment
  Change from baseline in the relative power spectral density of the delta and theta bands in patients.
Changes in Symbol Digit Modalities Test (SDMT) | At 6,12,18,24 months after enrollment
  Change from baseline in Symbol Digit Modalities Test (SDMT, scores range from 0 to 110, with lower scores indicating more severe cognitive impairment).
Changes in Montreal Cognitive Assessment Test (MoCA) | At 6,12,18,24 months after enrollment
  Change from baseline in Montreal Cognitive Assessment Test (MoCA, scores range from 0 to 30, with lower scores indicating more severe cognitive impairment).
changes in Mini-Mental Status Exam (MMSE) | At 6,12,18,24 months after enrollment
  Change from baseline in Mini-Mental Status Exam (MMSE, scores range from 0 to 30, with lower scores indicating more severe cognitive impairment.)

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital ,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang M, Han J, Xia J, Lin M, Chen T, Ruan S, Wang Q, Men Y, Gao R, Zheng H, Li J, Qi Y, Chen S, Wang Y, Tang Y, Li D, Yang X, Qiu Z, Liu Z, Dong H, Zhao Y, Hao J. Chinese neuroimmunological disease (NIDBase) cohort study: cohort profile. BMJ Open. 2026 Jan 8;16(1):e099386. doi: 10.1136/bmjopen-2025-099386. PMID 41506767